CLINICAL TRIAL: NCT01300169
Title: A Randomized Clinical Trial of the Collaborative Assessment and Management of Suicidality Versus Enhanced Care as Usual for Suicidal Soldiers
Brief Title: Operation Worth Living Project With Suicidal Soldiers at Ft. Stewart
Acronym: OWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of America (Other)
Collaborators: University of Washington (Other); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, David A. Jobes, Ph.D., Professor of Psychology, The Catholic University of America
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CUA-001; 09134002 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Suicidal Ideation Active; Suicidal and Self-injurious Behavior
Keywords: Suicide; Assessment; Intervention; CAMS
MeSH Terms: conditions — Self-Injurious Behavior; Suicide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAMS--Collaborative Driver-Treatment (Experimental): The Collaborative Assessment and Management of Suicidality (CAMS) is a suicide-specific clinical intervention that targets and treats patient-defined suicidal "drivers" over the course of clinical care.
  Interventions: Behavioral: The Collaborative Assessment and Management of Suicidality
- Enhanced Care as Usual--E-CAU (Active Comparator): This control group treatment will reflect current clinical practices for treating suicidal soldiers in the research site setting. These are providers were on site clinicians who provided care according to their usual and customary practices for working with suicidal risk within outpatient care.
  Interventions: Behavioral: Enhanced Care as Usual

INTERVENTIONS:
Behavioral: The Collaborative Assessment and Management of Suicidality — Intensive outpatient, suicide-focused, psychotherapy designed to target and treat the "drivers" of suicidal ideation and behaviors.
  Arms: CAMS--Collaborative Driver-Treatment
Behavioral: Enhanced Care as Usual — This is just standard outpatient mental health care that is routinely provided in the study site outpatient clinic
  Arms: Enhanced Care as Usual--E-CAU

SUMMARY:
This is a randomized controlled trial comparing the use of new clinical intervention (the "Collaborative Assessment and Management of Suicidality--CAMS") versus enhanced care as usual for suicidal Soldiers who are seen at outpatient mental health clinics at Ft. Stewart GA.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial of 148 suicidal active-duty US Army Soldiers. Participants were randomized to on-site providers who were trained in the Collaborative Assessment and Management of Suicidality (CAMS) vs. providers doing their own routine care--referred to as Enhanced Care as Usual (E-CAU) within an outpatient military treatment center. The CAMS Rating Scale (CRS) was used to reliably verify fidelity between treatment conditions and the adherence by CAMS providers to the model. Participants received informed consent to be randomly assigned to treatment arm and were ask to complete study assessments at baseline, 3 months, 6 months, and 12 months after the start of treatment. Recruitment is complete and all study assessments were completed as of March 2016. The study is in a second year of no cost extension; outcome data analyses and moderator analyses are currently underway to develop manuscripts for submission to peer-review scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Active duty Army personnel at FSGA
* Significant suicidal ideation
* Soldier is appropriate under FSGA policies
* Consent at baseline and follow up
* Consent to randomization and being digitally recorded

Exclusion Criteria:

* Significant psychosis, cognitive or physical impairment to not give consent
* Judicially ordered treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Scale for Suicidal Ideation | Baseline, post-treatment, 1, 3, 6, 12 months
  Industry standard for self-report suicidal ideation

SECONDARY OUTCOMES:
Overall symptom distress | Baseline, post treatment, 1, 3, 6, 12 months
  Outcome Questionnaire-45

CONTACTS AND LOCATIONS:
Overall Officials: David A. Jobes, Ph.D., Principal Investigator — The Catholic University of America

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lynch T, Bathe VC, Jobes DA. The Content of Patient-Identified Suicidal Drivers within CAMS Treatment Planning. Arch Suicide Res. 2024 Jan-Mar;28(1):411-417. doi: 10.1080/13811118.2022.2151958. Epub 2022 Dec 22. PMID 36550770
- [Derived] Corona CD, Gutierrez PM, Wagner BM, Jobes DA. The psychometric properties of the Collaborative Assessment and Management of Suicidality rating scale. J Clin Psychol. 2019 Jan;75(1):190-201. doi: 10.1002/jclp.22699. Epub 2018 Oct 6. PMID 30291761
- [Derived] Jobes DA, Comtois KA, Gutierrez PM, Brenner LA, Huh D, Chalker SA, Ruhe G, Kerbrat AH, Atkins DC, Jennings K, Crumlish J, Corona CD, Connor SO, Hendricks KE, Schembari B, Singer B, Crow B. A Randomized Controlled Trial of the Collaborative Assessment and Management of Suicidality versus Enhanced Care as Usual With Suicidal Soldiers. Psychiatry. 2017 Winter;80(4):339-356. doi: 10.1080/00332747.2017.1354607. PMID 29466107